CLINICAL TRIAL: NCT01912495
Title: Efficacy of 12 Week Boceprevir in Addition to Standard of Care Therapy Consisting of Peginterferon-alpha-2b and Ribavirin for the Treatment of Acute HCV Genotype 1 in HIV Co-infected Patients. A Proof of Concept Feasibility Clinical Trial.
Brief Title: Dutch Acute HCV in HIV Study (DAHHS)
Acronym: DAHHS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Onze Lieve Vrouwe Gasthuis (Other); UMC Utrecht (Other); University Medical Center Groningen (Other); Maastricht University Medical Center (Other); Rijnstate Hospital (Other); Slotervaart Hospital (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Bart Rijnders, MD,PhD, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL44825.078.13
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatitis C; Human Immunodeficiency Virus
MeSH Terms: conditions — Hepatitis C; Acquired Immunodeficiency Syndrome | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Boceprevir, peginterferon ribavirin (Experimental): All patients were intended to be treated in the 12 week peginterferon, ribavirin and boceprevir arm.
  Interventions: Drug: Boceprevir

INTERVENTIONS:
Drug: Boceprevir
  Other Names: Victrelis

SUMMARY:
Prospective open label proof of concept feasibility interventional clinical trial in which 60 acute HCV genotype 1 patients co-infected with HIV will receive 12 weeks of boceprevir in addition to Standard Of Care Peginterferon + Ribavirin if they show a Rapid Viral Responds at week 4.

The primary hypothesis of this study is that the subset of patients with a Rapid Viral Responds after 4 weeks of triple therapy with boceprevir, peginterferon alpha-2b (P) and ribavirin (RVR4) can be successfully treated with a shorter 12-week triple therapy regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Documented recent HCV genotype 1 infection (≤26 weeks old at the time of the baseline visit) according to definition mentioned below.
2. Plan to start a Standard Of Care therapy for acute HCV consisting of 24 weeks of Peginterferon + Ribavirin. HCV RNA plasma viral load at screening >1000 IU/ml.
3. A previously performed HCV RNA plasma measurement can be used for screening if <4 weeks old.
4. On HAART at the time of screening.
5. Minimum age 18 years.

Exclusion Criteria:

1. Disallowed co-medication that cannot be stopped or replaced: Several potentially life-threatening drug-drug interactions (DDI) are possible when boceprevir is combined with other drugs. Therefore ALL co-medication, including over-the-counter drugs should be checked for potential DDI with DDI table in the Dutch summary of product characteristics (SPC, appendix A). If the co-medication is not mentioned in the SPC DDI table, www.HCV-druginteractions.org should be used.
2. Contraindications for the use of full dose of peginterferon alpha-2b or ribavirin: neutrophils <0,75×109/l or thrombocytes < 100.000×109/l or a Hb <6.2mmol/L, creatinine clearance <50ml/min).
3. History of liver cirrhosis or >F1 fibrosis on fibroscan. Inclusion of patients with a chronic well-controlled HBV (HBV-DNA below the limit of detection) with tenofovir, lamivudine or emtricitabine therapy is allowed if fibroscan excludes >F1 fibrosis. Fibroscan reports <2 years old can be used for screening. Fibroscan is not required for other patients at screening.
4. HAART was started <4 weeks before baseline visit.
5. Inability to switch to a HAART regimen consisting of 2 nucleoside/tide reverse transcriptase inhibitors + Raltegravir (Isentress®) 400mg BID or rilpivirine 25mg QD or atazanavir (Reyataz®) 300mg QD + ritonavir (Norvir®) 100mg QD.
6. Patient that virologically failed HAART in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-08; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Rijnders, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (9):
- Netherlands (9):
  - Erasmus MC, Rotterdam, South Holland
  - AMC, Amsterdam
  - OLVG, Amsterdam
  - Slotervaart, Amsterdam
  - Ziekenhuis Rijnstate, Arnhem
  - UMCG, Groningen
  - MUMC, Maastricht
  - Radboud UMCN, Nijmegen
  - UMCU, Utrecht

REFERENCES:
- [Derived] Popping S, Cuypers L, Claassen MAA, van den Berk GE, De Weggheleire A, Arends JE, Boerekamps A, Molenkamp R, Koopmans MPG, Verbon A, Boucher CAB, Rijnders B, van de Vijver DAMC. Persistent Transmission of HCV among Men Who Have Sex with Men despite Widespread Screening and Treatment with Direct-Acting Antivirals. Viruses. 2022 Sep 2;14(9):1953. doi: 10.3390/v14091953. PMID 36146760
- [Derived] Hullegie SJ, Claassen MA, van den Berk GE, van der Meer JT, Posthouwer D, Lauw FN, Leyten EM, Koopmans PP, Richter C, van Eeden A, Bierman WF, Newsum AM, Arends JE, Rijnders BJ. Boceprevir, peginterferon and ribavirin for acute hepatitis C in HIV infected patients. J Hepatol. 2016 Apr;64(4):807-12. doi: 10.1016/j.jhep.2015.12.004. Epub 2015 Dec 12. PMID 26689767

RESULTS

PARTICIPANT FLOW:
Groups:
- Boceprevir: 12 week Boceprevir, Peginterferon and Ribavirin in RVR4 group
Period: Overall Study
Arm/Group | Boceprevir
Started | 57 (8 patients had only screening visit, total enrollment: 65)
Completed | 57
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Boceprevir/Peginterferon/Ribavirin: Boceprevir with Peginterferon and Ribavirin
Arm/Group | Boceprevir/Peginterferon/Ribavirin
Number analyzed (Participants) | 57
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [34 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 57
Region of Enrollment [Number; unit: participants]
  Netherlands | 57

OUTCOME MEASURES:

1. Primary Outcome: Sustained Viral Response(SVR) 12 Weeks of Follow up After the End of All Therapy for the Rapid Viral Response at Week 4(RVR4) Population.
Description: The outcome is a number of the patients with an undetectable Hepatitis C Virus (HCV) RNA at week 4 that have an undetectable HCV RNA 12 weeks after end of treatment.
Time Frame: 12 weeks
Population: 41 patients had a RVR4
Measure: Number; unit: participants
Groups:
- Boceprevir, Peginterferon and Ribavirin: 12 week Boceprevir, Peginterferon and Ribavirin
Arm/Group | Boceprevir, Peginterferon and Ribavirin
Number analyzed (Participants) | 41
participants | 41

2. Secondary Outcome: SVR 12 Weeks After the End of All Therapy in the Entire Study Population (With or Without RVR4).
Description: The outcome is a number of all patients who started treatment having an undetectable HCV RNA 12 weeks after the end of therapy
Time Frame: 12 weeks
Population: Total intention to treat population
Measure: Number; unit: participants
Groups:
- Boceprevir, Peginterferon and Ribavirin: 12 week boceprevir, peginterferon and ribavirin in intention to treat group
Arm/Group | Boceprevir, Peginterferon and Ribavirin
Number analyzed (Participants) | 57
participants | 49

3. Secondary Outcome: SVR 12 Weeks After End of Therapy in Patients With Already a RVR at Week 1.
Description: The number of patients who were undetectable for HCV at week one that had an undetectable HCV RNA load 12 weeks after the end of treatment
Time Frame: 12 weeks
Population: All patients having a rapid viral response at week 4 had a sustained viral response at 12(SVR12) weeks after treatment.
Measure: Number; unit: participants
Arm/Group | Boceprevir, Peginterferon and Ribavirin
Number analyzed (Participants) | 5
participants | 5

4. Secondary Outcome: SVR 12 Weeks After End of Therapy in Patients That Started Therapy ≤12weeks After the Presumed HCV Infection Date Versus Those After 12 Weeks.
Description: The number of patients having a undetectable HCV RNA 12 weeks after the end of treatment in the group patients that was treated within 12 week of calculated transmission date.
Time Frame: 12 weeks
Population: 5 patients were treated within 12 weeks after calculated transmission date. All other patients were treated between 12 and 26 weeks after calculated transmission date.
Measure: Number; unit: participants
Groups:
- Boceprevir Peginterferon Ribavirin: 12 week Boceprevir peginterferon and ribavirin
Arm/Group | Boceprevir Peginterferon Ribavirin
Number analyzed (Participants) | 5
participants | 5

5. Secondary Outcome: Alterations of Biomarkers by Therapy Induced Viral Eradication: Viral Sequencing, Mutation Analysis, Gene Expression Analysis, and RNA Analysis.
Time Frame: 72 weeks
Population: data were not collected during this study
Groups:
- Boceprevir Peginterferon Ribavirin: Boceprevir peginterferon and ribavirin
Arm/Group | Boceprevir Peginterferon Ribavirin
Number analyzed (Participants) | 0

6. Secondary Outcome: Safety: Treatment Related (Serious) Adverse Events ((S)AE) and Treatment Discontinuation for (S)AE.
Description: only serious adverse events are recorded in this secondary endpoint
Time Frame: 72 weeks
Population: 57 patients started treatment and were at risk
Measure: Number; unit: participants
Arm/Group | Boceprevir, Peginterferon and Ribavirin
Number analyzed (Participants) | 57
participants | 3

ADVERSE EVENTS:
Arm/Group | Boceprevir
Serious Adverse Events (participants affected / at risk) | 3/57
Other Adverse Events (participants affected / at risk) | 54/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Boceprevir (N=57)
Myocardial infarction (Cardiac disorders) | 1 — One myocardial infarction in a patient with a high-grade left anterior descending artery stenosis that was stented uneventfully (hemoglobin (Hb) 8∙7 mmol/L at the time of the infarction).
transient ischemic attack (Vascular disorders) | 1 — One suspected transient ischemic attack that resolved spontaneously and with normal MRI findings (Hb 6∙6 mmol/L)
anemia (General disorders) | 1 — One anemia (Hb 5·1 mmol/L) for which a transfusion was given and the ribavirin dose was decreased.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Boceprevir (N=57)
Anemia (Blood and lymphatic system disorders) | 47 — Grade 1 anemia was observed in 83%
anemia (Blood and lymphatic system disorders) | 7 — grade 2 anemia was observed in 12%

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes